CLINICAL TRIAL: NCT03818230
Title: An Evaluation of the Psychological Impact of Early Phase Clinical Trials in Cancer Patients.
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Natalie Cook, Honorary Consultant in Medical Oncology, University of Manchester
Other Study IDs: NHS001389
Record Dates: First submitted 2019-01-17; First posted 2019-01-28 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Cancer; Depression; Anxiety; Hope; Psychological Distress
Keywords: Clinical trials; Early phase clinical trials; Experimental cancer medicine
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None (observational study) — None (observational study)

SUMMARY:
This is an exploratory prospective observational cohort study to establish the levels of psychological distress in early phase clinical trial patients and evaluate the psychological impact of early phase clinical trials on cancer patients. Participants will be requested to complete self-reported questionnaires, measuring levels of anxiety, depression and hope, at different time points along the clinical trials pathway.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Able to provide informed consent
* Are being considered for an early phase clinical trial

Exclusion Criteria:

* Patients unable to comprehend English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to the Experimental Cancer Medicine Team (ECMT) at The Christie NHS Foundation Trust, to be considered for participation in an early phase clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Levels of anxiety and depression as per the Hospital Anxiety and Depression Scale questionnaire. | Approximately 14 weeks.

SECONDARY OUTCOMES:
Levels of hope as per the Adult Hope Scale. | Approximately 14 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No